CLINICAL TRIAL: NCT03446508
Title: Investigating Multi-electrode tDCS in Improving Word Finding and Memory Retrieval in Individuals With Mild Cognitive Impairment
Brief Title: Investigating HD-tDCS in Improving Word Finding and Memory Retrieval in Individuals With MCI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Associate professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-21
Record Dates: First submitted 2018-01-22; First posted 2018-02-26 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Mild Cognitive Impairment
Keywords: High definition transcranial direct stimulation; Mild Cognitive Impairment; Memory
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active frontal (Experimental): Active HD-tDCS
  Interventions: Device: Active frontal
- Active parietal (Experimental): Active HD-tDCS
  Interventions: Device: Active parietal
- Sham control (Sham Comparator): Sham HD-tDCS
  Interventions: Device: Sham

INTERVENTIONS:
Device: Active frontal — 1) active HD-tDCS will be administered
  Arms: Active frontal
Device: Active parietal — 2) active HD-tDCS will be administered
  Arms: Active parietal
Device: Sham — 3) sham HD-tDCS - no current
  Arms: Sham control

SUMMARY:
This study is attempting to improve word finding and memory retrieval problems persons with mild cognitive impairment (MCI) may have.

DETAILED DESCRIPTION:
This study attempts to improve word finding and memory retrieval problems in persons with mild cognitive impairment (MCI). To remember and find words, the brain has to search for the correct memory and MCI can negatively affect this search. Studies have suggested that low level electrical stimulation of the memory retrieval circuit can improve memory recall. The purpose of this study is to find the exact influence of multi-electrode or High Definition transcranial Direct Current Stimulation (HD-tDCS) by targeting a frontal and a parietal brain area, and their roles in memory retrieval/word finding in MCI. By modulating ongoing activity in 6 sessions of HD-tDCS the study investigates whether HD-tDCS may be used as a way to improve memory retrieval/word finding evaluated by cognitive measures and electroencephalography (EEG) measures before the first session and after the last session of HD-tDCS with a follow-up session 1-month after the stimulation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 90
2. Capable of understanding and signing an informed consent
3. Experiencing severe memory problems

Exclusion Criteria:

1. Severe organic co-morbidity
2. Pace maker / defibrillator
3. Pregnancy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Memory retrieval/word finding assessment. | Baseline (before the first HD-tDCS session), immediate post (immediately after the last HD-tDCS session) and 1 month follow up (1 month after the last HD-tDCS session)
  Changes in cognitive performance are compared between the 3 groups to investigate the influence of HD-tDCS on memory retrieval/word finding.

SECONDARY OUTCOMES:
Electroencephalography (EEG). | Baseline (before the first HD-tDCS session), immediate post (immediately after the last HD-tDCS session) and 1 month follow up (1 month after the last HD-tDCS session)
  Brain activity is recorded with electroencephalography (EEG) and is compared between the 3 groups to investigate the influence of HD-tDCS on memory retrieval/word finding.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided